CLINICAL TRIAL: NCT04089735
Title: A Multicenter, Randomized, Double-Masked, Two-Part, Placebo-Controlled Phase 2A Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of APP13007 for the Treatment of Inflammation and Pain After Cataract Surgery
Brief Title: A Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of APP13007 to Treat Inflammation and Pain After Cataract Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Formosa Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPN-201
Record Dates: First submitted 2019-08-28; First posted 2019-09-13 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Ocular Inflammation and Pain After Cataract Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- APP13007 0.05% twice daily (BID) [Part A] (Experimental): 1 drop 0.05% APP13007 twice daily for 21 days to the operated eye
  Interventions: Drug: APP13007, 0.05%
- APP13007 0.05% Placebo twice daily (BID) [Part A] (Experimental): 1 drop matching vehicle placebo for 0.05% APP13007 twice daily for 21 days to the operated eye
  Interventions: Drug: APP13007 Placebo, 0.05%
- APP13007 0.05% twice daily (BID) and once daily (QD) [Part B] (Experimental): 1 drop 0.05% APP13007 twice daily for 3 days followed by 1 drop once daily for 11 days to the operated eye
  Interventions: Drug: APP13007, 0.05%
- APP13007 0.05% Placebo twice daily (BID) and once daily (QD) [Part B] (Experimental): 1 drop matching vehicle placebo for 0.05% APP13007 twice daily for 3 days followed by 1 drop once daily for 11 days to the operated eye
  Interventions: Drug: APP13007 Placebo, 0.05%
- APP13007 0.1% twice daily (BID) and once daily (QD) [Part B] (Experimental): 1 drop 0.1% APP13007 twice daily for 3 days followed by 1 drop once daily for 11 days to the operated eye
  Interventions: Drug: APP13007, 0.1%
- APP13007 0.1% Placebo twice daily (BID) and once daily (QD) [Part B] (Experimental): 1 drop matching vehicle placebo for 0.1% APP13007 twice daily for 3 days followed by 1 drop once daily for 11 days to the operated eye
  Interventions: Drug: APP13007 Placebo, 0.1%

INTERVENTIONS:
Drug: APP13007, 0.05% — APP13007 eye drop, 0.05%
  Arms: APP13007 0.05% twice daily (BID) [Part A]; APP13007 0.05% twice daily (BID) and once daily (QD) [Part B]
Drug: APP13007, 0.1% — APP13007 eye drop, 0.1%
  Arms: APP13007 0.1% twice daily (BID) and once daily (QD) [Part B]
Drug: APP13007 Placebo, 0.05% — APP13007 placebo eyedrop, 0.05%
  Arms: APP13007 0.05% Placebo twice daily (BID) [Part A]; APP13007 0.05% Placebo twice daily (BID) and once daily (QD) [Part B]
Drug: APP13007 Placebo, 0.1% — APP13007 placebo eyedrop, 0.1%
  Arms: APP13007 0.1% Placebo twice daily (BID) and once daily (QD) [Part B]

SUMMARY:
This is a Phase 2a, 2-part study (designated Parts A and B) that will evaluate APP13007 dose strength and dosing frequency in a randomized double-masked fashion for comparison to the respective matching vehicle placebo. Part A will be conducted first to evaluate 0.05% APP13007 and matching vehicle placebo in an approximate 1:1 ratio in approximately 42 subjects who experience postoperative inflammation on the first day following routine, uncomplicated, cataract surgery and who meet all eligibility criteria. Based on the results of Part A, Part B of the study may be open for enrollment to evaluate 0.05% and/or 0.1% APP13007 at various dosing frequency in approximately 84 subjects, also in an approximate 1:1 ratio, active vs. placebo. In each Part, subjects will return periodically for study assessments during the treatment period and then for a follow-up visit approximately 1 week after stopping the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Expected to undergo unilateral uncomplicated cataract extraction via phacoemulsification and posterior chamber intraocular lens implantation in one eye.
* In Investigator's opinion, have Early Treatment Diabetic Retinopathy Study estimated potential of 0.7 (20/100) or better in study eye.
* Have > 10 and ≤ 30 cells in anterior chamber.
* Have an intraocular pressure ≤ 30 mmHg.

Exclusion Criteria:

* Have an anterior chamber cell count > 0 or any evidence of intraocular inflammation.
* Have a score > 0 on Ocular Pain Assessment in either eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — AimMax Therapeutics Inc.
Locations (9):
- United States (9):
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - United Medical Research Institute, Inglewood, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Levenson Eye Associates, Jacksonville, Florida
  - Bowden Eye and Associates, Jacksonville, Florida
  - Ophthalmology Associates, St Louis, Missouri
  - Eye Care Specialists, Kingston, Pennsylvania
  - Keystone Research Ltd., Austin, Texas
  - Cataract & Glaucoma Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-center US study in which 9 sites recruited subjects between August 2019 and October 2019 for Study Part A and between November 2019 and February 2020 for Study Part B
Pre-assignment Details: Of 52 enrolled participants for Part A, 45 met inclusion criteria and were randomized to treatment. Of 113 enrolled participants for Part B, 87 met inclusion criteria and were randomized to treatment.
Groups:
- APP13007 0.05% Twice Daily (BID): 1 drop 0.05% APP13007 twice daily for 21 days to the operated eye
  APP13007, 0.05%: APP13007 eye drop, 0.05%
- APP13007 0.05% Placebo Twice Daily (BID): 1 drop matching vehicle placebo for 0.05% APP13007 twice daily for 21 days to the operated eye
  APP13007 Placebo, 0.05%: APP13007 placebo eyedrop, 0.05%
- APP13007 0.05% Twice Daily (BID) and Once Daily (QD): 1 drop 0.05% APP13007 twice daily followed by 1 drop once daily to the operated eye
  APP13007, 0.05%: APP13007 eye drop, 0.05%
- APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD): 1 drop matching vehicle placebo for 0.05% APP13007 twice daily followed by 1 drop once daily to the operated eye
  APP13007 Placebo, 0.05%: APP13007 placebo eyedrop, 0.05%
- APP13007 0.1% Twice Daily (BID) and Once Daily (QD): 1 drop 0.1% APP13007 twice daily followed by 1 drop once daily to the operated eye
  APP13007, 0.1%: APP13007 eye drop, 0.1%
- APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD): 1 drop matching vehicle placebo for 0.1% APP13007 twice daily followed by 1 drop once daily to the operated eye
  APP13007 Placebo, 0.1%: APP13007 placebo eyedrop, 0.1%
Period: Overall Study
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
Started | 22 | 23 | 22 | 22 | 22 | 21
Completed | 21 | 17 | 20 | 16 | 21 | 15
Not Completed | 1 | 6 | 2 | 6 | 1 | 6
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Rescue therapy, prohibited medication, withdrawn requiring alternate medication for inflammation | 0 | 3 | 0 | 5 | 1 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD) | Total
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 22 | 21 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (8.6) | 66.3 (6.6) | 66.8 (6.6) | 70.0 (5.0) | 70.0 (6.0) | 65.2 (6.3) | 67.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 16 | 14 | 16 | 9 | 87
  Male | 5 | 8 | 6 | 8 | 6 | 12 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 3 | 2 | 2 | 3 | 18
  Not Hispanic or Latino | 18 | 19 | 19 | 20 | 20 | 18 | 114
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 2 | 3 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 6 | 2 | 2 | 2 | 20
  White | 15 | 18 | 15 | 18 | 17 | 18 | 101
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 23 | 22 | 22 | 22 | 21 | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events
Description: Number of treatment emergent adverse events and number of participants.
Time Frame: From First dose to Post-operative Day 28 (Part A) or Day 22 (Part B)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 22 | 21
Participants | 4 | 7 | 3 | 8 | 6 | 3

2. Primary Outcome: Intraocular Pressure - Change From Baseline (POD1 Prior to Dosing) to End-of-Treatment in the Operated Study Eye
Description: Intraocular pressure is measured in mm Hg at each study visit with a Goldmann applanation tonometer. The change from baseline is calculated by subtracting the pretreatment measurement value from the value at each visit.
Time Frame: Baseline and Post-operative Day 22 (Part A) or Day 15 (Part B)
Population: Safety Population - Participants who had the IOP data at End of Treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
Number analyzed (Participants) | 20 | 16 | 19 | 16 | 20 | 15
mmHg | 1.1 (4.2) | -2.3 (4.0) | -2.37 (3.71) | -2.38 (3.14) | -1.28 (4.36) | -1.00 (2.30)

3. Primary Outcome: Absolute Anterior Chamber Cell Count - Change From Baseline (POD1 Prior to Dosing) to POD 15 in the Operated Study Eye
Description: The number of cells in the anterior chamber of the eye are counted using slit-lamp biomicroscopy at each study visit and the results are reported as number of cells in a 1mm x 1mm area.
Time Frame: Baseline and Post-operative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 22 | 21
cells/mm^2 | -16.64 (5.80) | -9.24 (10.34) | -11.48 (8.65) | -5.67 (11.73) | -11.90 (4.73) | -7.43 (11.15)

4. Primary Outcome: Visual Acuity - Change From Baseline (POD1 Prior to Dosing) to End-of Treatment in the Operated Study Eye
Description: The visual acuity in each eye is corrected using the pinhole method and the acuity is quantified on a logMAR (minimal angle of resolution) scale using the 'Early Treatment Diabetic Retinopathy Study' [ETDRS] charts for right and left eyes. A logMAR Score is calculated using the number of incorrect letters.
Time Frame: Baseline and Post-operative Day 22 (Part A) or Day 15 (Part B)
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: logMAR score
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 22 | 21
logMAR score | -0.179 (0.266) | -0.073 (0.174) | -0.106 (0.184) | -0.024 (0.133) | -0.130 (0.165) | -0.025 (0.192)

5. Primary Outcome: Ocular Pain Grade - Change From Baseline (POD1 Prior to Dosing) to POD15 in the Operated Study Eye
Description: Ocular pain is measured in each eye using a subject-reported five-point (0-4) ocular pain grade scale (0 = no pain; 4 = severe pain).
Time Frame: Baseline and Post-operative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: grade
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 22 | 21
grade | -0.8 (1.0) | -0.4 (1.1) | -1.1 (1.0) | -0.4 (2.0) | -0.6 (1.2) | -0.3 (1.5)

6. Secondary Outcome: Subjects With Anterior Chamber Cell Count = 0 at POD15 in the Operated Study Eye Without Rescue Medication
Description: as for outcome 3
Time Frame: Post-operative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 22 | 21
Participants | 15 | 8 | 10 | 7 | 13 | 8

7. Secondary Outcome: Subjects With Ocular Pain Grade = 0 at POD 15 in the Operated Study Eye Without Rescue Medication
Description: as for outcome 5
Time Frame: Post-operative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 22 | 21
Participants | 21 | 16 | 20 | 16 | 19 | 15

8. Secondary Outcome: Anterior Chamber Flare - Change From Baseline (POD1 Prior to Dosing) to End-of Treatment in the Operated Study Eye
Description: The degree of turbidity (flare) in the anterior chamber of the eye is measured using slit-lamp biomicroscopy and quantified on a five-point (0-4) anterior chamber flare grade scale (0 = none; 4 = Intense). The change from baseline is calculated by subtracting the pretreatment measurement value from the value at each visit.
Time Frame: Baseline and Post-operative Day 22 (Part A) or Day 15 (Part B)
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: grade
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 22 | 21
grade | -1.05 (0.58) | -0.39 (0.94) | -0.77 (0.81) | -0.48 (0.96) | -0.64 (0.49) | -0.10 (1.04)

9. Secondary Outcome: Subjects Using of Anti-inflammatory 'Rescue' Medication Through End-of-Treatment
Description: Subjects who do not respond to study treatment after randomization (anterior chamber cell count > 30 cells or an increase in anterior chamber cell count by > 15 cells from pre-dose baseline or ≥ 2 grade of increase in anterior chamber flare from pre-dose baseline) are started on anti-inflammatory medication (referred to as 'Rescue' medication). The number of subjects starting 'Rescue' medication is recorded at each study visit.
Time Frame: First dose to Post-operative Day 22 (Part A) or Day 15 (Part B)
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 22 | 21
Participants | 0 | 3 | 0 | 5 | 0 | 5

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from informed consent through Post-operative Day 28 for Study Part A and informed consent through Post-operative Day 22 for Study Part B. Other (not Including Serious) adverse events were collected from the first dose through Post-operative Day 28 for Study Part A; from the first dose through Post-operative Day 22 for Study Part B.
Arm/Group | APP13007 0.05% Twice Daily (BID) | APP13007 0.05% Placebo Twice Daily (BID) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/22 | 0/22 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/22 | 0/22 | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 2/22 | 6/23 | 2/22 | 5/22 | 1/22 | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APP13007 0.05% Twice Daily (BID) (N=22) | APP13007 0.05% Placebo Twice Daily (BID) (N=23) | APP13007 0.05% Twice Daily (BID) and Once Daily (QD) (N=22) | APP13007 0.05% Placebo Twice Daily (BID) and Once Daily (QD) (N=22) | APP13007 0.1% Twice Daily (BID) and Once Daily (QD) (N=22) | APP13007 0.1% Placebo Twice Daily (BID) and Once Daily (QD) (N=21)
Eye inflammation (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Exploratory Phase 2 study with small sample sizes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institutions and Investigators participating in this trial shall have no right to publish or present the results of this study without the prior written consent of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT04089735/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT04089735/SAP_001.pdf